CLINICAL TRIAL: NCT06985082
Title: Risk Factors for Postoperative Complications in Pediatric Cardiac Surgery: A Retrospective Observational Study
Brief Title: This is an Observational Study That Aims to Demonstrate Postoperative Risk Factors in Pediatric Cardiac Surgery
Acronym: PEDS-CARE
Status: Not yet recruiting | Type: Observational
Sponsor: Instituto de Cardiologia do Rio Grande do Sul (Other)
Responsible Party: Principal Investigator, Caroline Kirschen Bristot, Anesthesiologist, Instituto de Cardiologia do Rio Grande do Sul
Other Study IDs: 6166.25
Record Dates: First submitted 2025-05-07; First posted 2025-05-22 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Arrhythmia; Acute Kidney Injuries; Sepsis; Pneumopathy; Thrombosis; Ventricular Asynchrony in Cardiac Surgery Patients; Pediatric Cardiac Surgery
Keywords: Pediatric Cardiac Surgery; Risk Factors Postoperative; Complications Posoperative
MeSH Terms: conditions — Arrhythmias, Cardiac; Acute Kidney Injury; Sepsis; Lung Diseases; Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: THERE IS NOT A INTERVENTION — THERE IS NOT A INTERVENTION

SUMMARY:
This retrospective observational study aims to identify risk factors for postoperative complications in children undergoing cardiac surgery at a tertiary hospital in Brazil. By analyzing both electronic and physical medical records, researchers will examine demographic, clinical, surgical, and laboratory data, focusing on variables such as cardiopulmonary bypass (CPB) time, use of vasoactive drugs, and the occurrence of complications such as arrhythmias, acute kidney injury, and infections. Statistical analysis will include both descriptive and inferential methods, with multivariate logistic regression used to identify predictors of adverse outcomes. The study will be conducted between 2025 and 2027 with an estimated budget of R$1,000. Its goal is to inform preventive strategies and optimize perioperative care, ultimately improving patient outcomes and reducing hospital costs.

DETAILED DESCRIPTION:
Congenital heart disease (CHD) affects approximately 1% of births and, although surgical advances have significantly reduced mortality, postoperative complications still represent a major challenge. Cardiopulmonary bypass (CPB) has been associated with adverse outcomes, such as longer mechanical ventilation time, prolonged hospital stay and hospital infections, which reinforces the importance of identifying predictors of complications. In this context, this study seeks to analyze the main risk factors that influence the recovery of children undergoing cardiac surgeries, contributing to the improvement of perioperative management.

This is a retrospective observational study, which will be conducted based on the analysis of medical records of pediatric patients undergoing cardiac surgeries in a tertiary hospital in Brazil. The research will allow the evaluation of clinical, surgical and laboratory variables, aiming to identify patterns and associations between perioperative factors and postoperative complications. This approach is justified by the wide availability of data, allowing robust statistical analyses, in addition to enabling the identification of clinical trends relevant to medical practice.

The study's general objective is to identify risk factors for postoperative complications in pediatric cardiac surgeries. To this end, it seeks to evaluate the incidence and types of complications, analyze the relationship between extracorporeal circulation time and adverse outcomes, in addition to identifying perioperative variables associated with mortality, length of hospital stay and hospital costs.

Data collection will be performed retrospectively based on the analysis of electronic and physical medical records, ensuring patient confidentiality and anonymity. A standardized instrument will be used to extract information, covering demographic characteristics, preoperative information, intraoperative data, postoperative complications and clinical outcomes. Data collected include age, sex, weight, height, cardiac diagnosis, CPB time, and use of vasoactive drugs, in addition to the occurrence of complications such as arrhythmias, acute kidney injury, and hospital infections. Data storage and organization will follow strict security protocols, ensuring restricted access to the responsible researchers. The informed consent form will be waived.

Statistical analysis will be conducted using descriptive and inferential methods. Categorical variables will be expressed as frequencies and percentages, while continuous variables will be presented as means and standard deviations or medians and interquartile ranges, according to their distribution. Initially, comparisons between groups will be performed using appropriate statistical tests, such as the t-test, Mann-Whitney, chi-square, and Fisher's exact test. To identify predictive factors of postoperative complications, multivariate logistic regression will be applied, in addition to calculations of predictive performance, including ROC curve, sensitivity, and specificity. The results will be considered statistically significant for p < 0.05, and the analyses will be conducted using SPSS 25.0 and STATA 12.0 software.

The study will be conducted between 2025 and 2027, including submission to the Ethics Committee, data collection, statistical analysis and final defense. The total estimated budget for the research is R$ 1,000.00, covering costs for data collection materials, printing and acquisition of scientific literature.

Therefore, this study seeks to provide crucial information for reducing postoperative complications and optimizing care for pediatric patients undergoing cardiac surgeries. The identification of predictive factors will allow the development of preventive strategies and more effective interventions, contributing to improving the quality of life of these patients and reducing hospital costs.

ELIGIBILITY:
Inclusion Criteria:

* All patients under 18 years of age who underwent cardiac surgery

Exclusion Criteria:

* Patients undergoing non-cardiac thoracic surgeries
* Patients over 18 years of age
* Pregnant women will be excluded from the study

Max Age: 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: Children under 18 years of age undergoing elective or emergency pediatric cardiac surgeries, performed with or without extracorporeal circulation, will be included.
Sampling Method: Probability Sample
Enrollment: 310 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2025-05 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Risk Factors | 2 years
  To identify risk factors associated with postoperative complications in pediatric cardiac surgeries performed in a tertiary hospital in Brazil.

SECONDARY OUTCOMES:
The Incidence | 2 years
  To assess the incidence and types of cardiac and extracardiac complications after pediatric cardiac surgery.
CPB and Complications | 2 years
  Analyze the relationship between duration of extracorporeal circulation and postoperative complications.
Adverse Outcomes | 2 years
  Identify perioperative risk factors associated with adverse outcomes
The influence of complications | 2 years
  Analyze how postoperative complications influence length of hospital stay, mortality and hospital costs

IPD SHARING:
Plan to Share IPD: Undecided